CLINICAL TRIAL: NCT01979198
Title: Thoracolumbar Burst Fracture Treated With Pedicle Screws: Radiographic Analysis of Discs and Vertebral Body Height at Fractured and Adjacent Levels
Brief Title: Thoracolumbar Burst Fracture Treated With Pedicle Screws: Radiographic Outcomes
Status: Completed | Type: Observational
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, Chief, Division of Spine Surgery, Dep. of Orthopedics and Traumatology, Taipei Veterans General Hospital, Taiwan
Other Study IDs: 2012-03-030BC
Record Dates: First submitted 2013-10-16; First posted 2013-11-08 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-10

CONDITIONS: Burst Fracture
Keywords: burst fracture, kyphotic angle, surgical outcome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- fusion group: close reduction with posterior short-segment transpedicular screw fixation with posterior fusion
- non-fusion group: close reduction with posterior short-segment transpedicular screw fixation without posterior fusion

SUMMARY:
The surgical results of thoracolumbar and lumbar burst fracture have been reported to be comparable between patients with and without fusion in a midterm follow-up. There is, however, no report comparing the results of fusion and non-fusion with a long-term follow-up. Therefore, a long term comparative study is still needed to focus on the issues of functional and radiographic outcomes, especially preservation of the motion segment in the long run, to determine whether fusion should be a routine procedure for surgically treated burst fractures of the thoracolumbar and lumbar spines. Therefore, we report herein a long-term comparative study of fusion and non-fusion based on our previous work, with an average 134 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* neurologically intact spine with a kyphotic angle more than 20o, decreased vertebral body height more than 50% or a canal compromise more than 50%;
* incomplete neurological deficit with a canal compromise less than 50%;
* complete neurological deficit;
* multilevel spinal injury or multiple trauma.

Exclusion Criteria:

* progression of the neurological deficit;
* a canal compromise still more than 50% in those who showed no improvement of the neurological deficit.

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients suffered from burst fracture of the thoracolumbar and lumbar spine
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2012-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Radiologic outcomes | postoperative 6 weeks
  * Injured vertebral body height
  * Kyphotic angle
  * Regional segmental motion
Radiologic outcomes | postoperative 12 weeks
  * Injured vertebral body height
  * Kyphotic angle
  * Regional segmental motion
Radiologic outcomes | postoperative 6 months
  * Injured vertebral body height
  * Kyphotic angle
  * Regional segmental motion
Radiologic outcomes | postoperative 12 months
  * Injured vertebral body height
  * Kyphotic angle
  * Regional segmental motion
Radiologic outcomes | postoperative 24 months
  * Injured vertebral body height
  * Kyphotic angle
  * Regional segmental motion
Radiologic outcomes | up to postoperative 161 months
  * Injured vertebral body height
  * Kyphotic angle
  * Regional segmental motion

SECONDARY OUTCOMES:
Functional outcomes | postoperative 24 months
  * Greenough Low Back Outcome Scale
  * Visual Analogue Scale (VAS) for back pain
  * Neurologic status: Frankel grading system
Functional outcomes | up to postoperative 161 months
  * Greenough Low Back Outcome Scale
  * Visual Analogue Scale (VAS) for back pain
  * Neurologic status: Frankel grading system

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Tien Wang, MD, Principal Investigator — Department of Orthopedics and Traumatology, Taipei Veterans General Hospital
Locations (1):
- Dep. of Orthopedics and Traumatology, Taipei Veterans General Hospital, Taipei, Taiwan